CLINICAL TRIAL: NCT03363958
Title: Effect of Remote Ischemic Conditioning on Ischemia and Reperfusion Injury in Patients Submitted to Coronary Artery Bypass Grafting.
Brief Title: Remote Ischemic Conditioning to Attenuate Myocardial Death and Improve Operative Outcome.
Acronym: RICARDO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medinet Heart Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIPC Trial
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Coronary Artery Bypass; Myocardial Reperfusion Injur; Ischemic Preconditioning, Myocardial; Ischemic Postconditioning
Keywords: myocardial protection; remote ischemic preconditioning; remote ischemic postconditioning; cardiac surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC Group (Experimental): Three cycles of remote ischemic conditioning (5minutes ischemia and 5minutes reperfusion; lower leg ischemia achieved by pressure cuff inflation and deflation); First three cycles the patient will receive 24 hours preoperatively, second three cycles the patient will receive after the induction of general anesthesia but before skin incision shortly before CABG. Remote ischemic postconditioning (5minutes ischemia and 5minutes reperfusion; lower leg ischemia achieved by pressure cuff inflation and deflation) will be administered to the patient within 60 minutes after the completion of all coronary artery bypass grafts and the restoration of coronary blood flow.
  Interventions: Procedure: Remote Ischemic Preconditioning with Postconditioning
- Control Group (Sham Comparator): Control group will receive sham procedure near identical to intervention. That will be afforded by inflation of pressure cuff on artificial leg hidden under the draping by an assistant who is not included in the research team and does not have any connection to study design and data analysis.
  Interventions: Procedure: Sham RIPC procedure

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning with Postconditioning — Three cycles of 5 minutes of ischemia and 5 minutes of reperfusion of lower leg 24 hours, immediately before surgery and within 60 minutes after the restoration of coronary blood flow postoperatively.
  Arms: RIC Group
Procedure: Sham RIPC procedure — Three cycles of 5 minutes of inflation and 5 minutes of deflation of artificial lower leg immediately before surgery and within 60 minutes after the restoration of coronary blood flow postoperatively.
  Arms: Control Group

SUMMARY:
This study evaluates the addition of remote ischemic preconditioning and postconditioning to standard myocardial protection protocol in patients submitted to off - pump coronary artery bypass grafting in a prospective, 1:1 randomized, double blind fashion. An interventional group will receive remote ischemic preconditioning 24-hours before OP-CABG, immediately before surgery and within 60 minutes following surgery by means of lower limb ischemia achieved by pressure cuff inflation, whereas control group will receive sham procedure perioperatively.

DETAILED DESCRIPTION:
In a prospective, 1:1 randomized and double blind fashion, the study will evaluate the impact of remote ischemic preconditioning, both immediate and second window of protection (24 hours and immediately before surgery) with remote ischemic postconditiong on operative outcomes in patients submitted to coronary artery bypass grafting without use of extracorporeal circulation.

Remote ischemic conditioning was found to provide protection against necrosis and apoptosis due to ischemia and reperfusion injury, a phenomenon observed during coronary artery bypass grafting. That in turn was associated with poor postoperative outcomes, predominantly poor survival.

Remote ischemic preconditioning will be provided by repeated lower leg ischemia and reperfusion with pressure cuff inflation for five minutes and deflation for five minutes in three consecutive cycles. Remote ischemic preconditioning will be performed 24 hours before CABG and immediately before surgery. Remote ischemic postconditioning will be performed within 60 minutes following the last coronary artery bypass graft completion and the restoration of coronary blood flow.

The study will assess clinical endpoints such as postoperative acute myocardial infarction (type 5 MI), postoperative mortality, postoperative renal failure and laboratory outcomes such as postoperative serial measurements of troponin T release or glomerular filtration rate as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients qualified to coronary artery bypass grafting according to ESC/EACTS Guidelines of myocardial revascularization, suffering from:

* Multivessel coronary artery disease amenable for surgical treatment
* Negative history of previous cardiac or vascular surgery in childhood and afterwards.
* Negative history of active neoplastic disease, neither past medical history of oncological treatment
* Patients with non insulin dependent diabetes mellitus treated chronically with oral derivatives of sulfonylourea such as but not limited to: glibenclamide.

Exclusion Criteria:

Patients suffering from acute insuficiency of any organ/ system and those suffering from end stage organ failure such as:

* Chronic renal disease - KDOQI stage ≥ 3;
* Chronic renal failure class A by Child - Pugh'a;
* Chronic respiratory failure (type I and II according to Campbell et al. and type I according to Wood et al.);
* Chronic intermittent claudication class 2A according to Fontaine;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative myocardial necrosis | 72 hours postoperatively
  Serial mesurements of High - Sensitive Troponin T release
Postoperative kidney injury | 7 days postoperatively
  Serial measurements of estimated glomerular filtration rate by creatinine

SECONDARY OUTCOMES:
Perioperative mortality | 30 days postoperatively
  30-day all cause mortality
Perioperative myocardial infarction | 30 days postoperatively
  30-day myocardial infarction
Postoperative Acute Kidney Injury | 30 days
  Prevalence of acute kidney injury according to Society of Thoracic Surgeons definitions of outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub S. Marczak, M.D., Principal Investigator — Medinet Heart Center
Locations (1):
- Medinet Heart Centre, Nowa Sól, Lubusz Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marczak J, Nowicki R, Kulbacka J, Saczko J. Is remote ischaemic preconditioning of benefit to patients undergoing cardiac surgery? Interact Cardiovasc Thorac Surg. 2012 May;14(5):634-9. doi: 10.1093/icvts/ivr123. Epub 2012 Jan 26. PMID 22286602
- See also: Related Info — http://medinet.pl